CLINICAL TRIAL: NCT00254293
Title: A Study to Assess the Steady-State Trough Serum Concentration, Safety, and Immunogenicity of Abatacept (BMS-188667) Administered Subcutaneously in Subjects With Active Rheumatoid Arthritis Who Are Receiving Disease Modifying Ant-Rheumatic Drugs (DMARDs)
Brief Title: Study to Assess Steady-State Trough Concentrations, Safety, and Immunogenicity of Abatacept After Subcutaneous (SC) Administration to Subjects With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-063
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Group 1 (weight < 60 kg) (Placebo Comparator)
  Interventions: Drug: Abatacept or Placebo (both as IV & SC Solution)
- Group 2 (weight < 60 kg) (Placebo Comparator)
  Interventions: Drug: Abatacept or Placebo (both as IV & SC Solution)
- Group 3 (weight 60-100 kg) (Placebo Comparator)
  Interventions: Drug: Abatacept or Placebo (both as IV & SC solution)
- Group 4 (weight > 100 kg) (Placebo Comparator)
  Interventions: Drug: Abatacept or Placebo (both as IV & SC solution)
- Group 5 (weight > 100 kg) (Placebo Comparator)
  Interventions: Drug: Abatacept or Placebo (both as IV & SC solution)
- Abatacept (Experimental): Long Term
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept or Placebo (both as IV & SC Solution) — Abatacept & Placebo as IV & SC solution, IV/SC, Abatacept 500 mg IV (Day 1)/Abatacept 75 mg SC (once weekly for 12 weeks) or Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks), 12 weeks then long term extension (LTE).
  Other Names: Orencia
  Arms: Group 1 (weight < 60 kg)
Drug: Abatacept or Placebo (both as IV & SC Solution) — Abatacept & Placebo as IV & SC solution, IV/SC, Abatacept 500 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks), 12 weeks then long term extension (LTE).
  Other Names: Orencia
  Arms: Group 2 (weight < 60 kg)
Drug: Abatacept or Placebo (both as IV & SC solution) — Abatacept & Placebo as IV & SC solution, IV/SC, Abatacept 750 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks), 12 weeks then long term extension (LTE).
  Other Names: Orencia
  Arms: Group 3 (weight 60-100 kg)
Drug: Abatacept or Placebo (both as IV & SC solution) — Abatacept & Placebo as IV & SC solution, IV/SC, Abatacept 1000 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks), 12 weeks then long term extension (LTE).
  Other Names: Orencia
  Arms: Group 4 (weight > 100 kg)
Drug: Abatacept or Placebo (both as IV & SC solution) — Abatacept & Placebo as IV & SC solution, IV/SC, Abatacept 1000 mg IV (Day 1)/Abatacept 200 mg SC (once weekly for 12 weeks) or Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks), 12 weeks then long term extension (LTE).
  Other Names: Orencia
  Arms: Group 5 (weight > 100 kg)
Drug: Abatacept — Solution in pre-filled syringes, Subcutaneously, 125 mg, Weekly
  Arms: Abatacept

SUMMARY:
The purpose of this study is to study serum levels of Abatacept after subcutaneous dosing in subjects with RA.

ELIGIBILITY:
Inclusion Criteria:

* Meet ARA criteria for diagnosis of RA with active disease.
* RA diagnosis for at least 1 year.
* > = 6 swollen joints.
* > = 8 tender joints.
* Taking methotrexate (MTX) or MTX plus not more than 1 added oral DMARD for > = 3 months and stable for 28 days prior to dosing.

Exclusion Criteria:

* Serious acute or bacterial infection in last 3 months.
* Chronic or recurrent bacterial infections.
* History of TB within previous 3 years or old TB not adequately treated.
* Specific lab test abnormalities
* History of cancer within 5 years.
* Exposure to CTLA4Ig (Cytotoxic T-lymphocyte (T-cell)-associated antigen 4Ig), belatacept, rituximab, efalizumab, alefacept, or other investigational drug or biologic.
* Treatment with hydroxychloroquine, azathioprine, leflunomide, immunoadsorption columns, mycophenolate mofetil, cyclosporine, D-Penicillamine or calcineurin inhibitors.
* Exposure to live vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-01; Primary Completion 2007-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Orlando Clinical Research Center, Orlando, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - New Orleans Center For Clinical Research, New Orleans, Louisiana
  - Davita Clinical Research, Minneapolis, Minnesota
  - The Arthritis Clinic & Carolina Bone & Joint, Charlotte, North Carolina

REFERENCES:
- [Derived] Westhovens R, Kremer JM, Moreland LW, Emery P, Russell AS, Li T, Aranda R, Becker JC, Qi K, Dougados M. Safety and efficacy of the selective costimulation modulator abatacept in patients with rheumatoid arthritis receiving background methotrexate: a 5-year extended phase IIB study. J Rheumatol. 2009 Apr;36(4):736-42. doi: 10.3899/jrheum.080813. Epub 2009 Feb 27. PMID 19273451
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Short term (12 week) randomized Period: started January 2006/completed May 2007. Long term extension (LTE): started April 2006/completed July 2012. During LTE: variable dose period and fixed dose period. Patients with active Rheumatoid Arthritis (RA) and receiving disease modifying anti-rheumatic drugs (DMARDS) were eligible to participate.
Pre-assignment Details: Enrolled/not treated (19): prior treatment not washed out; no longer met study criteria; withdrew consent before treatment. To enter LTE, participant completed the short term period, and was assigned to a variable SC dose group (75, 125, 200 mg SC abatacept) based on body weight; completers of variable dose LTE rolled over into fixed dose LTE.
Groups:
- Group 1: 500 mg IV/75 mg SC: Short term (ST) randomized 12 week period: Abatacept or Placebo as intravenous (IV) and subcutaneous (SC) administration: Abatacept 500 mg IV (Day 1)/Abatacept 75 mg SC (once weekly for 12 weeks); body weight < 60 kg. Long term extension (LTE) variable dosing period: 75 mg abatacept SC administered weekly following an IV loading dose (IV abatacept for participants randomized to placebo in ST period, loading dose as described in group 1 description, or IV placebo for participants randomized to abatacept in ST period) on Day 85 (IV abatacept based on their weight at screening; < 60 kg received 500 mg abatacept IV, 60 - 100 kg received 750 mg abatacept IV, > 100 kg received 1000 mg abatacept IV for participants randomized to placebo in ST period)or, IV placebo for participants randomized to abatacept in ST period). At Day 365(1-year anniversary visit), subjects were reweighed for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
- Group 2: 500 mg IV/125 mg SC: Short term (ST) randomized 12 week period: Abatacept 500 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo;body weight < 60 kg. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period; loading dose described in Group 1 description, or IV placebo for participants randomized to abatacept in ST period). Variable Long term for 125 mg SC: body weight <60 to >100 kg. Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
- Group 3 : 750 mg IV/125 mg SC: Short term (ST) randomized 12 week period: Abatacept 750 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo (body weight 60-100 kg). Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose described in Group 1 description, or IV placebo for participants randomized to abatacept in ST period). Variable Long term for 125 mg SC: body weight <60 to >100 kg). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Group 4: 1000mg IV/125 mg SC: Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo; Body weight > 100 kg. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose as described in group 1 description, or IV placebo for participants randomized to abatacept in ST period); variable long term for 125 mg SC: body weight <60 to >100 kg) . Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Group 5: 1000 mg IV/200 mg SC: Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 200 mg SC (once weekly for 12 weeks) or Placebo; body weight > 100 kg. Long term extension (LTE) variable dosing period: 200 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose based on weight as described in Group 1 description, or IV placebo for participants randomized to abatacept in ST period). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
- Placebo: Short term (ST) randomized 12 week period: Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks), by body weight. Long term extension (LTE) variable dosing period: all placebo participants rolled over to a variable dose of abatacept SC (75, 125, 200 mg) administered weekly following an IV loading dose of abatacept on Day 85. Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
- Fixed Dose 125 mg Abatacept: Participants who completed the variable dose long term extension (LTE)period and received variable doses of subcutaneous (SC) abatacept (75, 125, 200 mg SC) were rolled over into the LTE with fixed dose, irrespective of body weight: SC abatacept 125 milligram (mg) in pre-filled syringes, administered Weekly.
Period: Short Term (12 Week) Randomized Dosing
Arm/Group | Group 1: 500 mg IV/75 mg SC | Group 2: 500 mg IV/125 mg SC | Group 3 : 750 mg IV/125 mg SC | Group 4: 1000mg IV/125 mg SC | Group 5: 1000 mg IV/200 mg SC | Placebo | Fixed Dose 125 mg Abatacept
Started | 7 | 4 | 29 | 6 | 5 | 17 (2, 2, 9, 2, and 2 were randomized to placebo in body weight Groups 1, 2, 3, 4, 5, respectively.) | 0
Completed | 7 | 3 | 26 | 5 | 5 | 17 | 0
Not Completed | 0 | 1 | 3 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — poor/non-compliance by participant | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: LTE Open Label Variable SC Dosing
Arm/Group | Group 1: 500 mg IV/75 mg SC | Group 2: 500 mg IV/125 mg SC | Group 3 : 750 mg IV/125 mg SC | Group 4: 1000mg IV/125 mg SC | Group 5: 1000 mg IV/200 mg SC | Placebo | Fixed Dose 125 mg Abatacept
Started | 11 (Participants who received ST placebo rolled over to 75mg SC dose group (by body weight, <60kg).) | 0 (Participants rolled over to 125mg dose group summarized as one group (body weight <60 to >100 kg).) | 42 (Variable SC dose group: 125 mg Weekly, body weight <60 to >100kg (Groups 2, 3, 4 in ST Period).) | 0 (Participants rolled over to 125mg dose group summarized as one group (body weight <60 to >100 kg).) | 10 (Participants who received ST placebo rolled over to variable SC dose group (by body weight, >100kg).) | 0 (Participants rolled over to a variable SC dose group of 75, 125 or 200 mg Weekly by body weight.) | 0 (Participant rolled over from LTE (Variable Dose Period) to LTE (Fixed Dose Period).)
Completed | 8 | 0 | 32 | 0 | 8 | 0 | 0
Not Completed | 3 | 0 | 10 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Poor or non-compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: LTE Open Label Fixed Dosing
Arm/Group | Group 1: 500 mg IV/75 mg SC | Group 2: 500 mg IV/125 mg SC | Group 3 : 750 mg IV/125 mg SC | Group 4: 1000mg IV/125 mg SC | Group 5: 1000 mg IV/200 mg SC | Placebo | Fixed Dose 125 mg Abatacept
Started | 0 | 0 | 0 | 0 | 0 | 0 | 48
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 35
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 13
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Poor or non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline includes all participants enrolled and treated. Baseline parameters are presented for each arm but the total value for baseline mean age and standard deviation (SD) includes all participants in LTE. Data are presented by treatment the participant actually received, not to what they were randomized to receive.
Groups:
- Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg): Short term (ST) randomized 12 week period: Abatacept or Placebo as intravenous (IV) and subcutaneous (SC) administration: Abatacept 500 mg IV (Day 1)/Abatacept 75 mg SC (once weekly for 12 weeks); Long term extension (LTE) variable dosing period: 75 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, IV placebo for participants randomized to abatacept in ST period).
- Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg): Short term (ST) randomized 12 week period: Abatacept 500 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, IV placebo for participants randomized to abatacept in ST period).
- Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg): Short term (ST) randomized 12 week period: Abatacept 750 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 ((IV abatacept for participants randomized to placebo in ST period, IV placebo for participants randomized to abatacept in ST period). Participants from Group 3 in ST period were rolled into Group 2 for LTE variable dosing period (125 mg SC abatacept).
- Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg): Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, IV placebo for participants randomized to abatacept in ST period). Participants from Group 4 in ST period were rolled into Group 2 for LTE variable dosing period (125 mg SC abatacept).
- Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg): Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 200 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 200 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, IV placebo for participants randomized to abatacept in ST period).
- Placebo: Short term (ST) randomized 12 week period: Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks). Long term extension (LTE) variable dosing period: all placebo participants were rolled over to a variable dose of abatacept SC administered weekly following an IV loading dose of abatacept on Day 85.
- Total: Total of all reporting groups
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo | Total
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (5) | 64 (10) | 59 (12) | 51 (9) | 55 (9) | 59 (11) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 26 | 5 | 4 | 12 | 57
  Male | 0 | 1 | 3 | 1 | 1 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 29 | 6 | 5 | 17 | 68

OUTCOME MEASURES:

1. Primary Outcome: Short Term Period: Steady-state Trough Serum Concentration (Cmin) of Abatacept Following Weekly Subcutaneous Dosing in Participants With Active Rheumatoid Arthritis Receiving Disease Modifying Anti-rheumatic Drugs (DMARDS)
Description: Participants received abatacept while also receiving DMARDS over a short term (ST) 12 Week period. To eliminate contribution from the IV loading dose of abatacept during the short term study period, Cmin values were selected from Days 71 to 85, when contribution from IV was negligible. Minimum trough serum concentration of abatacept (Cmin) was measured in micrograms/milliliter (µg/mL). Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Days 71 to 85
Population: 50 of the 51 abatacept-treated subjects were included. One subject who discontinued after receiving only Day 1 dosing was not included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg): Subjects randomized to abatacept in group 1 received an intravenous (IV) loading dose of abatacept on Day 1 of 500 mg followed by 75 mg subcutaneous (SC) abatacept (once weekly for 12 weeks).
- Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg): Subjects randomized to abatacept in group 2 received an intravenous (IV) loading dose of abatacept on Day 1 of 500 mg followed by 125 mg subcutaneous (SC) abatacept (once weekly for 12 weeks).
- Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg): Subjects randomized to abatacept in group 3 received an intravenous (IV) loading dose of abatacept on Day 1 of 750 mg followed by 125 mg subcutaneous (SC) abatacept (once weekly for 12 weeks).
- Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg): Subjects randomized to abatacept in group 4 received an intravenous (IV) loading dose of abatacept on Day 1 of 1000 mg followed by 125 mg subcutaneous (SC) abatacept (once weekly for 12 weeks).
- Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg): Subjects randomized to abatacept in group 5 received an intravenous (IV) loading dose of abatacept on Day 1 of 1000 mg followed by 200 mg subcutaneous (SC) abatacept (once weekly for 12 weeks).
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg)
Number analyzed (Participants) | 7 | 4 | 29 | 5 | 5
µg/mL
  Day 71 | 22.64 (20.13) | 28.03 (42.13) | 24.05 (40.65) | 16.22 (24.39) | 26.52 (56.53)
  Day 78 | 21.66 (19.99) | 34.17 (29.49) | 24.41 (52.35) | 11.57 (32.25) | 29.21 (52.96)
  Day 85 | 23.62 (31.63) | 36.73 (31.64) | 24.93 (38.42) | 13.01 (41.35) | 27.53 (58.87)

2. Secondary Outcome: Short Term Period: Peak Serum Concentration (Cmax) of Abatacept at Steady State in Participants With Rheumatoid Arthritis Receiving DMARDS
Description: Peak serum concentration (Cmax) of abatacept after weekly SC administration was determined between the SC dosing interval from Day 71 to 78. Abatacept in human serum was measured by enzyme-linked immunosorbent assay (ELISA). Lower limit of quantification (LLOQ) was 0.001, Upper limit of quantification (ULOQ) was 0.030. Cmax measured in micrograms per milliliter(µg/mL). Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 71 to Day 78
Population: Pharmacokinetic (PK) analysis set included those participants treated with abatacept and having PK data available
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg)
Number analyzed (Participants) | 7 | 4 | 26 | 5 | 5
µg/mL | 26.3 (29.5) | 34.9 (46.6) | 31.9 (42.8) | 14.7 (44.3) | 41.7 (41.2)

3. Secondary Outcome: Short Term Period: Area Under the Curve (AUC) in Time Interval of 7 Days [AUC(TAU)] of Abatacept in Participants With Rheumatoid Arthritis Receiving DMARDS
Description: The steady-state pharmacokinetic parameter AUC(TAU) of abatacept after weekly SC administration was determined between the SC dosing interval from Day 71 to 78 (TAU=7 days). Abatacept in human serum was measured by enzyme-linked immunosorbent assay (ELISA). Lower limit of quantification (LLOQ) was 0.001; Upper limit of quantification (ULOQ) was 0.030. AUC(TAU) measured in in micrograms*hours per milliliter (µg*h/mL). Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 71 to Day 78
Population: Pharmacokinetic (PK) analysis set included those participants treated with abatacept and having PK data available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg)
Number analyzed (Participants) | 7 | 3 | 24 | 4 | 5
µg*h/mL | 4066 (22.2) | 6699 (20.7) | 4607 (38.6) | 2555 (30.1) | 5849 (40.5)

4. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, Discontinuations Due to Adverse Events Reported During the Variable Dosing Phase of the Long Term Period (LTE)
Description: AEs during variable dose phase of LTE + 56 days post last dose in the variable dose phase or start of the fixed dose phase, which ever came first; includes deaths reported during the variable dose phase including those that occurred greater than 56 days after last dose. Medical Dictionary for Regulatory Activities (MedDRA) version: 15.1. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization (included hospitalizations for elective surgical procedures). Treatment-related=having certain, probable, possible, or missing relationship to study drug. Data presented by treatment the participant was randomized to and not what they actually received.
Time Frame: Day 85 to 56 days post last dose
Population: Participants included those that rolled over into the LTE, receiving variable SC dosing of abatacept in the Variable Dose Period.
Measure: Number; unit: participants
Groups:
- 75 mg SC Abatacept (Body Weight < 60 kg): Long term extension (LTE) variable dosing period: 75 mg abatacept SC administered weekly following an IV loading dose (IV abatacept for participants randomized to placebo in ST period, loading dose 500 mg IV (Day 1)/Abatacept 75 mg SC (once weekly), or IV placebo for participants randomized to abatacept in ST period) on Day 85 (IV abatacept based on their weight at screening; < 60 kg received 500 mg abatacept IV, 60 - 100 kg received 750 mg abatacept IV, > 100 kg received 1000 mg abatacept IV for participants randomized to placebo in ST period)or, IV placebo for participants randomized to abatacept in ST period). At Day 365(1-year anniversary visit), subjects were reweighed for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
- 125 mg SC Abatacept (Body Weight <60 to >100 kg): Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose (IV abatacept for participants randomized to placebo in ST period, or IV placebo for participants randomized to abatacept in ST period) on Day 85 (IV abatacept based on their weight at screening; < 60 kg received 500 mg abatacept IV, 60 - 100 kg received 750 mg abatacept IV, > 100 kg received 1000 mg abatacept IV for participants randomized to placebo in ST period)or, IV placebo for participants randomized to abatacept in ST period). At Day 365(1-year anniversary visit), subjects were reweighed for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- 200 mg SC Abatacept (Body Weight > 100 kg): 200 mg abatacept SC administered weekly following an IV loading dose on Day 85 (1000 mg IV abatacept for participants randomized to placebo in ST period, or IV placebo for participants randomized to abatacept in ST period). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
Arm/Group | 75 mg SC Abatacept (Body Weight < 60 kg) | 125 mg SC Abatacept (Body Weight <60 to >100 kg) | 200 mg SC Abatacept (Body Weight > 100 kg)
Number analyzed (Participants) | 11 | 42 | 10
participants
  Deaths | 0 | 1 | 0
  Participants with SAEs | 2 | 13 | 4
  Participants with drug related SAEs | 1 | 2 | 1
  Participants discontinued due to SAEs | 0 | 1 | 1
  Participants with AEs | 9 | 38 | 9
  Participants with drug related AEs | 2 | 20 | 3
  Participants discontinued due to AEs | 1 | 2 | 1

5. Secondary Outcome: Short Term Period: Summary of Adverse Events (AEs), Serious AEs, Deaths, and Discontinuations Due to AEs During 12 Weeks of Treatment With Either Abatacept or Placebo
Description: Number of Participants with Adverse events (AEs), Serious AEs, discontinuations due to AEs, or Deaths occurring while participant was on treatment from Day 1 (treatment) to Day 85 or early termination from the study. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization (also included hospitalizations for elective surgical procedures). Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 1 to Day 85 (or early termination)
Measure: Number; unit: participants
Groups:
- Placebo (by Body Weight Category): Subjects randomized to placebo in the ST period received IV placebo followed by SC placebo (once weekly for 12 weeks).
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17
participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Participants with SAEs | 0 | 1 | 1 | 0 | 1 | 0
  Participants with AEs | 5 | 3 | 21 | 6 | 5 | 11
  Discontinued due to AEs | 0 | 1 | 0 | 1 | 0 | 0

6. Secondary Outcome: Short Term Period: Number of Participants With Pre-specified Adverse Events (AEs) of Special Interest After Administration of Abatacept or Placebo Over 12 Weeks
Description: AEs of special interest: infection and/or infestation; neoplasms (benign, malignant, unspecified; autoimmune disorder; infusional AEs (peri-infusional: AEs occurring during first 24 hours (hrs) after start of the IV loading dose; acute infusional: AEs occurring during the first hour after the start of the IV loading dose; injection site AEs: AEs occurring at the site of the SC injection. Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 1 to Day 85 (or early termination)
Population: All subjects treated were analyzed for safety.
Measure: Number; unit: participants
Groups:
- Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg): Subjects randomized to abatacept in group 1 received an IV loading dose of abatacept on Day 1 of 500 mg followed by abatacept 75 mg SC (once weekly for 12 weeks).
- Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg): Subjects randomized to abatacept in group 2 received an IV loading dose of abatacept on Day 1 of 500 mg followed by abatacept 125 mg SC (once weekly for 12 weeks).
- Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg): Subjects randomized to abatacept in group 3 received an IV loading dose of abatacept on Day 1 of 750 mg followed by abatacept 125 mg SC (once weekly for 12 weeks).
- Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg): Subjects randomized to abatacept in group 4 received an IV loading dose of abatacept on Day 1 of 1000 mg followed by abatacept 125 mg SC (once weekly for 12 weeks).
- Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg): Subjects randomized to abatacept in group 5 received an IV loading dose of abatacept on Day 1 of 1000 mg followed by abatacept 200 mg SC (once weekly for 12 weeks).
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17
participants
  Number with Infection/Infestation events | 3 | 1 | 9 | 3 | 1 | 4
  Number with malignant neoplasm events | 0 | 0 | 0 | 0 | 0 | 0
  Number with autoimmune disorder events | 0 | 0 | 0 | 0 | 0 | 0
  Number with acute infusional events | 0 | 0 | 2 | 1 | 0 | 0
  Number with peri-infusional events | 0 | 0 | 4 | 3 | 0 | 0
  General disorders and injection site events | 0 | 1 | 11 | 3 | 2 | 1

7. Secondary Outcome: Short Term Period: Mean Percent Change From Baseline on Day 85 in Participants Positive for Serum Rheumatoid Factor During Abatacept or Placebo Administration
Description: Serum samples were obtained on Days 1, 8, 15, 29, 57 and day of discharge (Day 85 or earlier) for determination of presence of rheumatoid factor (RF). Baseline was defined as Day 1 to calculate percent change. Lower limit of quantitation (LLQ) was 5 Units/milliliter (U/mL). Values below LLQ were set to 2.5 U/mL. Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 1 to Day 85 (or early termination)
Population: Analysis set included all available data from participants who received abatacept or placebo. For RF analysis in Group 1 Day 1/Day 85 number of participants = 7/7; Group 2 = 3/3; Group 3 = 29/29; Group 4 = 6/6; Group 5 = 5/5; Placebo = 17/15 participants.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Groups:
- Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg): Short term (ST) 12 week period: Abatacept as intravenous (IV) and subcutaneous (SC) administration: Abatacept 500 mg IV (Day 1)/Abatacept 75 mg SC (once weekly for 12 weeks).
- Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg): Short term (ST) 12 week period: Abatacept 500 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks).
- Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg): Short term (ST) randomized 12 week period: Abatacept 750 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks).
- Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg): Short term (ST) 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks).
- Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg): Short term (ST) 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 200 mg SC (once weekly for 12 weeks).
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 3 | 29 | 6 | 5 | 15
percentage of change from baseline | -1.50 (43.50) | -8.89 (3.14) | -17.69 (26.61) | -16.29 (16.24) | -19.32 (15.21) | 43.72 (154.47)

8. Secondary Outcome: Short Term Period: Number of Participants With Laboratory Abnormalities in Hematology at Baseline (Day 1) to End of Period (Day 85)
Description: Blood samples were obtained: At screening, within 24 hours prior to study drug administration on Day 1, on Days 15, 29, 57 and at study discharge. Baseline (BL) defined as Day 1 prior to treatment. Common toxicity criteria (CTC), Version 3 used to assess parameters. lower limit of normal (LLN). ANC=absolute neutrophil count. White blood cells Grade (Gr) 1:<LLN to 3.0*10^9/L, Gr 2:<3.0 to 2.0*10^9/L, Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L. ANC Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Lymphocytes Gr 1: <LLN to 3.0, Gr 2: 2.0 < 3.0, Gr 3: 1.0 to < 2.0, Gr 4; < 1.0. Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Hematocrit (%): <0.75*pre-treatment. Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 1 to Day 85 (or early termination)
Population: All participants treated with either abatacept or placebo. Participant counted once in total for each arm but participant could have multiple AEs of different grade. Grade category is number of participants with that Grade of AE (Grades 1, 2, 3, 4)
Measure: Number; unit: participants
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17
participants
  Baseline (Day 1 prior to treatment) Total | 4 | 3 | 15 | 1 | 2 | 9
  Grade 1 baseline | 4 | 3 | 13 | 1 | 2 | 8
  Grade 2 baseline | 0 | 1 | 2 | 0 | 0 | 3
  Grade 3 baseline | 0 | 0 | 1 | 0 | 0 | 0
  Grade 4 baseline | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 after treatment to Day 85 Total | 4 | 4 | 20 | 1 | 4 | 13
  Grade 1 on treatment | 4 | 4 | 17 | 1 | 3 | 11
  Grade 2 on treatment | 0 | 1 | 6 | 0 | 1 | 3
  Grade 3 on treatment | 0 | 0 | 0 | 0 | 0 | 1
  Grade 4 on treatment | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Short Term Period: Number of Participants With Laboratory Abnormalities in Serum Chemistry at Baseline and on Treatment up to Day 85
Description: Screening, BL, Days 15, 29, 57, 85 or discharge. Upper limit of normal (ULN). CTC grade (Gr): Alanine transaminase Gr 1:>ULN to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Aspartate aminotransferase Gr 1: >ULN to 2.5*ULN; Gr 2:>2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. G-Glutamyl Transferase (U/L) Gr 1:>ULN to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Alkaline phosphatase (U/L) Gr 1:>ULN to 2.5*ULN, Gr2:>2.5 to 5.0*ULN, Gr3:>5.0 to 20.0*ULN, Gr4: >20.0*ULN; creatinine (mg/dL) Gr 1: >ULN to 1.5*ULN; Gr 2: >1.5 to 3.0*ULN; Gr 3: >3.0 to 6.0*ULN; Gr 4: >10.0*ULN. Albumin (g/dL) Gr 1:<LLN to 3.0; Gr 2:<3.0 to 2.0; Gr 3: <2.0. Uric Acid (mg/dL)Gr 1: >1.0 x ULN to 10.0; Gr 4: >10.0. Sodium (mEq/L) Gr 1: >ULN to 150; Gr 2: >150 to 155; Gr 3: >155 to 160; Gr 4: > 160. Potassium (mEq/L) Gr 1: >ULN to 5.5; Gr 2: >5.5 to 6.0; Gr 3: >6.0 to 7.0; Gr 4: >7.0. Data presented by treatment participant actually received.
Time Frame: Day 1 to Day 85 (or early termination)
Population: All participants treated with abatacept or placebo in the short term period. Participant is counted once in total but could have multiple AEs of different grade. Grade category is number of participants with that Grade of AE (Grades 1, 2, 3, 4)
Measure: Number; unit: participants
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17
participants
  Baseline (Day 1 prior to treatment) Total | 2 | 2 | 6 | 1 | 4 | 7
  Grade 1 baseline | 2 | 2 | 5 | 1 | 4 | 7
  Grade 2 baseline | 0 | 0 | 1 | 0 | 0 | 2
  Grade 3 baseline | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 baseline | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 (after treatment) to Day 85 Total | 5 | 4 | 18 | 3 | 4 | 15
  Grade 1 on treatment | 5 | 0 | 18 | 3 | 3 | 15
  Grade 2 on treatment | 1 | 0 | 4 | 0 | 0 | 4
  Grade 3 on treatment | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 on treatment | 0 | 0 | 0 | 0 | 1 | 0

10. Secondary Outcome: Short Term Period: Mean Change From Baseline at Day 85 in Blood Pressure After SC Administration of Abatacept or Placebo in Participants With Rheumatoid Arthritis Receiving DMARDS
Description: Blood pressure (systolic and diastolic) was recorded while the participant was seated during the screening visit, at baseline on Day 1 (prior to administration of IV infusion), prior to administration of all SC injections, and at study discharge (Day 85 or 7 days after the last dose for subjects who terminated early). In addition, blood pressure was recorded at 30 and 60 minutes after the start of the IV infusion on Day 1, and 30 and 60 minutes after all SC injections. Blood pressure was measured in millimeters of mercury (mm Hg). Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 1 to Day 85 (or early termination)
Population: All participants who were treated with abatacept or placebo and had vital signs taken were analyzed throughout the 12 weeks. At Day 85 N = 6, 3, 28,6, 5, 17 in groups 1, 2, 3, 4, 5, Placebo, respectively
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17
mm Hg
  Change from baseline in Diastolic blood pressure | -5.2 (10.0) | 0.0 (13.1) | 0.7 (7.5) | 3.5 (11.2) | -5.4 (9.6) | 1.8 (8.3)
  Change from baseline in Systolic blood pressure | -4.0 (12.1) | -6.3 (6.8) | 0.3 (17.8) | -0.8 (8.2) | -4.2 (10.5) | 0.2 (12.1)

11. Secondary Outcome: Short Term Period: Mean Change From Baseline at Day 85 in Pulse Rate After SC Administration of Abatacept or Placebo in Participants With Rheumatoid Arthritis Receiving DMARDS
Description: Pulse rate was taken while participant was seated. Pulse rate was recorded during the screening visit, at baseline on Day 1 (prior to administration of IV infusion), prior to administration of all SC injections, and at study discharge (Day 85 or 7 days after the last dose for subjects who terminated early). In addition, vital signs were recorded at 30 and 60 minutes after the start of the IV infusion on Day 1, and 30 and 60 minutes after all SC injections. Pulse rate measured in beats/min (bpm). Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Day 1 to Day 85 (or early termination)
Population: All participants who were treated with abatacept or placebo and had vital signs taken were analyzed throughout the 12 weeks. At Day 85 N = 6, 3, 28, 6, 5, 17 in groups 1, 2, 3, 4, 5, Placebo, respectively
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | Placebo (by Body Weight Category)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 17
bpm | -2.9 (10.0) | 0.3 (11.1) | -0.6 (9.5) | 3.5 (10.5) | -11.4 (9.0) | -1.0 (7.1)

12. Secondary Outcome: Short Term Period: Mean Change From Screening to Day 85 in Electrocardiogram (QT, PR Intervals, QRS Width) After SC Administration of Abatacept or Placebo in Participants With Rheumatoid Arthritis Receiving DMARDS
Description: A 12-lead electrocardiogram (ECG) was recorded at screening and at discharge from the study (Day 85 or 7 days after the last dose of study drug for those subjects who terminated early). If there was no history of known cardiac events, an ECG was performed within 6 months of study entry, and documentation was on file, then the screening ECG was not repeated at screening. QT interval, PR interval and QRW Width were reported in milliseconds (msec). If no ECG issues were found in the 12 weeks of the Short Term Period, ECG was not repeated during LTE. Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Screening to Day 85 (or early termination)
Population: A total of 68 participants were treated with abatacept or placebo: 66 had results at screening and 52 had results at Discharge (Day 85) for QT interval and QRS Width; 65 and 51 participants had PR interval results at Screening and Discharge (Day 85), respectively.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- All Treated Participants: ECG change from screening after treatment were summarized for all participants treated with either abatacept or placebo in the Short Term Period.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 66
msec
  Change from Screening in QT interval (N=52) | -1.47 (24.72)
  Change from Screening in PR interval (N=51) | 5.28 (21.10)
  Change from Screening in QRS Width (N=52) | 0.22 (11.03)

13. Primary Outcome: Number of Participants With Pre-specified AEs of Special Interest in the Variable Dosing Phase of Long Term Extension (LTE)
Description: LTE period with variable abatacept dosing starting on Day 85 and continuing until Day 533 when LTE fixed dosing started. AEs of special interest: infection and/or infestation; neoplasms (malignant); pre-specified autoimmune disorder; infusional AEs (peri-infusional: pre-specified AEs occurring during first 24 hours (hrs) after start of the IV loading dose; acute infusional: pre-specified AEs occurring during the first hour after the start of the IV loading dose; systemic injection site reactions (SIR): pre-specified AEs for SIR; local injection site reaction: pre-specified AEs for local site reaction. Data are presented by treatment the participant was randomized to and not what they actually received.
Time Frame: Day 85 to Day 533
Population: All 63 participants who completed the ST period enrolled into the LTE variable dosing period and were analyzed.
Measure: Number; unit: participants
Groups:
- 75 mg SC Abatacept: variable dosing period: 75 mg abatacept SC administered weekly following an IV loading dose (IV abatacept for participants randomized to placebo in ST period, or IV placebo for participants randomized to abatacept in ST period); body weight <60kg. At Day 365(1-year anniversary visit), subjects were reweighed for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
- 125 mg SC Abatacept: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose as described in group 1 description, or IV placebo for participants randomized to abatacept in ST period). Body weight <60 to >100 kg. Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- 200 mg SC Abatacept: 200 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, or IV placebo for participants randomized to abatacept in ST period); body weight >100kg. Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period
Arm/Group | 75 mg SC Abatacept | 125 mg SC Abatacept | 200 mg SC Abatacept
Number analyzed (Participants) | 11 | 42 | 10
participants
  Number with Serious Infection/Infestation | 1 | 1 | 2
  Number with Malignant Neoplasms | 1 | 5 | 1
  Number with Autoimmune Disorder | 0 | 1 | 0
  Number with Acute Infusional Event | 0 | 0 | 0
  Number with Serious Systemic injection Reaction | 0 | 0 | 0
  Number with Local Injection Site Reaction | 0 | 4 | 0

14. Secondary Outcome: Short Term Period: Mean Change From Screening at Day 85 in ECG (Heart Rate) After SC Administration of Abatacept or Placebo in Participants With Rheumatoid Arthritis Receiving DMARDS
Description: A 12-lead electrocardiogram (ECG) was recorded at screening and at discharge from the study (Day 85 or 7 days after the last dose of study drug for those subjects who terminated early). If there was no history of known cardiac events, an ECG was performed within 6 months of study entry, and documentation was on file, then the screening ECG was not repeated at screening. Heart Rate was reported in beats per minute (bpm). In no ECG issues were found in the 12 weeks of the Short Term Period, ECG was not repeated during LTE. Data are presented by treatment the participant actually received, not by what they were randomized to receive.
Time Frame: Screening to Day 85 (or early termination)
Population: A total of 68 participants were treated with abatacept or placebo: 65 had results at screening and 53 had results at Discharge (Day 85) for Heart Rate.
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- All Treated Participants: ECG Heart Rate change from screening after treatment were summarized for all participants treated with either abatacept or placebo in the Short Term Period
Arm/Group | All Treated Participants
Number analyzed (Participants) | 53
bpm | 0.51 (8.43)

15. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, Discontinuations Due to Adverse Events Summarized Over the Entire Long Term Extension (LTE) Period (Both Variable and Fixed Dosing)
Description: On Day 85 participants rolled over into the LTE with variable dose phase first and at Day 533, a fixed dose phase of 125 mg abatacept SC weekly, irrespective of body weight. This summary includes AEs reported during entire LTE treatment plus 56 days post last dose; includes all deaths reported during the LTE including those that occurred greater than 56 days after last dose. MedDRA version: 15.1. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization (also included hospitalizations for elective surgical procedures). Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Day 533 to 56 Days Post last dose
Population: total number of participants in the Long Term Extension Period.
Measure: Number; unit: participants
Groups:
- SC Abatacept: Overall summary of all participants in the LTE. LTE Period consisted of a variable dose (75 mg, 125 mg, 200 mg abatacept) phase first and at Day 533, a fixed dose phase of 125 mg abatacept SC weekly, irrespective of body weight.
Arm/Group | SC Abatacept
Number analyzed (Participants) | 63
participants
  Deaths | 6
  Participants with SAEs | 35
  Participants with Drug Related SAEs | 7
  Participants Discontinued due to SAEs | 3
  Participants with AEs | 61
  Participants with Drug Related AEs | 34
  Participants Discontinued due to AEs | 5

16. Secondary Outcome: Overall Study ST and LTE Periods: Number of Participants With Anti-abatacept Antibodies and/or Anti-cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Antibodies
Description: Assessment of positive antibody response based upon analysis using a validated enzyme-linked immunosorbent assay (ELISA) with a cut-off value. CTLA4 is a protein receptor that downregulates the immune system. Short Term (ST) period was initial 12 Weeks of the study. Overall LTE includes both the variable and fixed abatacept dosing periods and was from the end of the ST period (Day 85) up to 168 days post last dose (treatment in LTE ranged from 4.4 to 74.2 months. Data in the ST period are summarized by the treatment the participants actually received, while the LT period data are summarized by treatment the participant was randomized to receive.
Time Frame: ST: Day 1 to Day 85; LTE: Day 85 to 168 days post last dose
Population: In the ST period, only subjects treated with abatacept (51) were evaluated for antibodies. In LTE, 61 participants were analyzed for anti-abatacept antibodies, and 62 participants were analyzed for CTLA4-T antibodies. Participants were analyzed during treatment and post-treatment (28, 56, 85, and 168 days post-treatment).
Measure: Number; unit: participants
Groups:
- Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg): Short term (ST) 12 week period: Abatacept 750 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks).
- Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg): Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks).
- LTE (Variable and Fixed Dosing Abatacept): Long term extension (LTE) consisted of 2 periods: variable dosing of abatacept combined with DMARDS and fixed dosing abatacept combined with DMARDS. Participants were weighed prior to starting LTE (variable dosing) and dosing was assigned per body weight category. Variable dosing period required an IV loading dose prior to starting SC dosing (if participant had been randomized to placebo in the short term period). Variable dosing: 500 mg IV/75 mg SC and 500 mg IV/125 mg SC in participants less than (<)60 kg body weight; 750 mg IV/125 mg SC in participants between 60 and 100 kg body weight; 1000 mg IV/125 mg SC and 1000 mg IV/200 mg SC in participants greater than (>) 100 kg body weight. Participants were rolled over into a fixed SC dose of 125 mg per week in the fixed dosing period prior to their Year 2 anniversary visit for the study (as early as Day 533).
Arm/Group | Group 1: 500 mg IV/75 mg SC (Body Weight < 60 kg) | Group 2: 500 mg IV/125 mg SC (Body Weight < 60 kg) | Group 3 : 750 mg IV/125 mg SC (Body Weight 60-100 kg) | Group 4: 1000mg IV/125 mg SC (Body Weight > 100 kg) | Group 5: 1000 mg IV/200 mg SC (Body Weight > 100 kg) | LTE (Variable and Fixed Dosing Abatacept)
Number analyzed (Participants) | 7 | 4 | 29 | 6 | 5 | 62
participants
  Number with anti-abatacept antibodies | 0 | 0 | 0 | 1 | 0 | 11
  Number with anti-CTLA4 antibodies | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 of short term study up to 71 months in the long term study.
Description: AEs and SAEs are summarized by the treatment arm to which the participants were randomized.
Groups:
- Abatacept 1000mg IV/125mg SC: Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose as described in group 1 description, or IV placebo for participants randomized to abatacept in ST period). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Abatacept 1000mg IV/200mg SC: Short term (ST) randomized 12 week period: Abatacept 1000 mg IV (Day 1)/Abatacept 200 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 200 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose based on weight as described in Group 1 description, or IV placebo for participants randomized to abatacept in ST period). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Abatacept 500mg IV/125mg SC: Short term (ST) randomized 12 week period: Abatacept 500 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period; loading dose described in Group 1 description, or IV placebo for participants randomized to abatacept in ST period). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Abatacept 500mg IV/75mg SC: Short term (ST) randomized 12 week period: Abatacept or Placebo as intravenous (IV) and subcutaneous (SC) administration: Abatacept 500 mg IV (Day 1)/Abatacept 75 mg SC (once weekly for 12 weeks); Long term extension (LTE) variable dosing period: 75 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept based on their weight at screening; < 60 kg received 500 mg abatacept IV, 60 - 100 kg received 750 mg abatacept IV, > 100 kg received 1000 mg abatacept IV for participants randomized to placebo in ST period)or, IV placebo for participants randomized to abatacept in ST period). At Day 365(1-year anniversary visit), subjects were reweighed for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Abatacept 750mg IV/125mg SC: Short term (ST) randomized 12 week period: Abatacept 750 mg IV (Day 1)/Abatacept 125 mg SC (once weekly for 12 weeks) or Placebo. Long term extension (LTE) variable dosing period: 125 mg abatacept SC administered weekly following an IV loading dose on Day 85 (IV abatacept for participants randomized to placebo in ST period, loading dose described in Group 1 description, or IV placebo for participants randomized to abatacept in ST period). Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
- Abatacept (LT) 125 mg SC: Participants who completed the long term extension (LTE)period and received variable doses of subcutaneous (SC) abatacept (as described in Groups 1 - 5) were rolled over into the LTE with fixed dose: SC abatacept 125 milligram (mg) in pre-filled syringes, administered Weekly.
- Placebo (ST): Short term (ST) randomized 12 week period: Placebo IV(Day 1)/Placebo SC (once weekly for 12 weeks). Long term extension (LTE) variable dosing period: all placebo participants rolled over to a variable dose of abatacept SC (75, 125, 200 mg) administered weekly following an IV loading dose of abatacept on Day 85. Participants reweighed at 1 year anniversary for subsequent dosing to verify correct dosing in the variable-dose phase of the LTE period.
Arm/Group | Abatacept 1000mg IV/125mg SC | Abatacept 1000mg IV/200mg SC | Abatacept 500mg IV/125mg SC | Abatacept 500mg IV/75mg SC | Abatacept 750mg IV/125mg SC | Abatacept (LT) 125 mg SC | Placebo (ST)
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5 | 1/5 | 0/6 | 1/28 | 35/63 | 0/18
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 2/5 | 5/6 | 18/28 | 58/63 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 1000mg IV/125mg SC (N=6) | Abatacept 1000mg IV/200mg SC (N=5) | Abatacept 500mg IV/125mg SC (N=5) | Abatacept 500mg IV/75mg SC (N=6) | Abatacept 750mg IV/125mg SC (N=28) | Abatacept (LT) 125 mg SC (N=63) | Placebo (ST) (N=18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 7 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 1000mg IV/125mg SC (N=6) | Abatacept 1000mg IV/200mg SC (N=5) | Abatacept 500mg IV/125mg SC (N=5) | Abatacept 500mg IV/75mg SC (N=6) | Abatacept 750mg IV/125mg SC (N=28) | Abatacept (LT) 125 mg SC (N=63) | Placebo (ST) (N=18)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 13 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 3 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 7 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 3 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 5 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 14 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 14 | 3
Chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 13 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 7 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 4 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 4 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 5 | 3
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 11 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 7 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 10 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 5 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 8 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Headache (Nervous system disorders) | 3 | 2 | 0 | 0 | 1 | 8 | 3
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 6 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0 | 0 | 12 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 22 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 4 | 13 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 7 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 7 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1
Injection site swelling (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 8 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 5 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 4 | 0

LIMITATIONS AND CAVEATS:
Error resulted in 4 participants being treated with study drug they were not randomized to receive. ST data were summarized by study drug participants actually received while LT data were summarized by what participants were randomized to receive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.